CLINICAL TRIAL: NCT01999946
Title: Extended-Release Naltrexone Opioid Treatment at Jail Re-Entry
Acronym: XOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Friends Research Institute, Inc. (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03724; 1U01DA033336-01A1 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Heroin Dependence; Opioid-Related Disorders
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Extended-Release Naltrexone (XR-NTX) (Experimental): Extended-Release Naltrexone (Vivitrol®), 380mg administered 1x/month by intramuscular injection.
  Interventions: Drug: Extended-Release Naltrexone
- Enhanced Treatment As Usual (ETAU) (No Intervention): Enhanced Treatment As Usual arm will not receive any study medication, but will receive enhancement counseling centered on post-release treatment involvement and a patient-drug educational handout with direct referrals to re-entry community treatment, including agonist maintenance (methadone and buprenorphine programs), drug-free outpatient and 12-step resources, and residential treatment including supportive housing programs will be provided. These counseling and referral efforts are designed to exceed standard, out-of-treatment experiences, and will ensure both arms are offered tangible health benefits above and beyond that of the usual jail incarceration period in accordance with DHS prisoner research standards.
- Methadone Treatment Program (MTP) (No Intervention): Quasi-Experimental cohort, will be participants recruited from NYC Rikers Island jail's Key Extended Entry Program (KEEP)'s jail methadone maintenance program, they will not receive any intervention from study, but will receive enhancement counseling centered on post-release treatment involvement and a patient-drug educational handout with direct referrals to re-entry community treatment.These counseling and referral efforts are designed to exceed standard, out-of-treatment experiences, and will ensure both arms are offered tangible health benefits above and beyond that of the usual jail incarceration period in accordance with DHS prisoner research standards. MTP participants are new KEEP methadone participants not enrolled in community methadone at the time of arrest.

INTERVENTIONS:
Drug: Extended-Release Naltrexone — Extended-Release Naltrexone (Vivitrol®), 380mg administered 1x/month by intramuscular injection.
  Other Names: Vivitrol; XR-NTX
  Arms: Extended-Release Naltrexone (XR-NTX)

SUMMARY:
The purpose of this study is to compare the effectiveness of extended-release naltrexone (XR-NTX) vs. enhanced treatment-as-usual (TAU) among opioid dependent adults leaving NYC jails. In parallel, we propose to recruit a matched, quasi-experimental methadone cohort, which will result in a naturalistic comparison of XR-NTX vs. an established jail-based methadone treatment program standard-of-care. Our primary aim is to compare time-to-relapse among participants treated with XR-NTX vs. randomized TAU controls and time-to-relapse among XR-NTX arm vs. jail-based MTP participants, following release from jail. Secondary aims will compare related opioid treatment outcomes post-release across all arms.

DETAILED DESCRIPTION:
This study is a randomized control trial of XR-NTX (n=85) vs. enhanced TAU (n=85) among opioid dependent adults leaving NYC jails who explicitly reject agonist treatment. Initiating treatment the week prior to release and continuing for 24 weeks post-release, we hypothesize the XR-NTX arm will demonstrate significantly longer time-to-relapse vs. TAU. In parallel, we propose to recruit a matched, quasi-experimental methadone cohort (n=85), which will result in a naturalistic comparison of XR-NTX vs. an established jail-based MTP standard-of-care.

Rationale: Immediate relapse to drug, alcohol, and tobacco use is a nearly universal and expected near-term outcome among adults with addiction disorders leaving U.S. jails. Yet while opioid agonist therapies are proven and effective re-entry interventions, many US correctional facilities, including almost all large U.S. municipal jails, do not offer these treatments. However, in New York City (NYC), jail-to-community methadone treatment is, since 1986, a well-studied standard-of-care, yet many inmates eligible to initiate the methadone treatment program (MTP) while incarcerated do not, possibly due to anti-methadone patient preferences. Rather, the vast majority of these jail detainees undergo a brief 6-day methadone taper following arrest, remain in jail for brief periods out-of-treatment while 'drug free' and undergoing a decline in physiologic opioid tolerance, nearly universally relapse to heroin or other illicit opioid use following release, and are re-arrested in the next 12 months at rates of 50-75%. Extended-release naltrexone (XR-NTX, Vivitrol), now FDA-approved for opioid dependence, produces a 30-day mu opioid receptor antagonist blockade, and offers an potentially promising modality for 'inoculating' persons leaving jails against immediate opioid relapse. Persons injected with 380mg of XR-NTX are unable to effectively experience euphoria or respiratory depression when returning to average doses of illicit opioids for the ensuing 4-5 weeks. An injection prior to release would possibly give the individual a month or so to return home from jail, experience opioid abstinence, and then either continue XR-NTX, initiate agonist or behavioral treatments, or, resume a significantly postponed relapse to illicit use. Our team recently established the feasibility of administering XR-NTX to opioid dependent adults within a week of release in NYC jails. We now propose to conduct a large, definitive randomized controlled trial estimating the effectiveness of XR-NTX as opioid treatment at release from jail vs. a counseling- and referral-enhanced treatment-as-usual (TAU) condition. We also propose to recruit a non-randomized, quasi-experimental cohort of participants in a jail-based methadone maintenance program (MTP), allowing an additional comparison of XR-NTX to a methadone standard-of-care.

Specific Aim 1: Randomized Effectiveness Trial of XR-NTX vs. TAU for Jail-to-Community Re-Entry Opioid Relapse Prevention. Our primary aim is to compare time-to-relapse among participants treated with XR-NTX vs. randomized TAU controls, following release from jail.

Specific Aim 2: Quasi-Experimental Comparison of XR-NTX vs. a Methadone Treatment Program for Re-Entry Opioid Relapse Prevention. To compare time-to-relapse among the XR-NTX RCT arm vs. jail-based MTP participants using a quasi-experimental design.

Specific Aim 3a-e: Related Opioid Treatment Outcomes. To compare re-entry rates of 5 treatment outcomes across all arms: 3a) community treatment initiation and retention, 3b) any opioid and other illicit drug or alcohol use, defined as continuous counts of both days, amount/day, and urine toxicologies, 3c) injection drug use and HIV sexual risk factors, 3d) accidental drug overdose and mortality, and, 3e) rates of re-incarceration and an exploratory analysis of cost-effectiveness.

Implications: While there is growing interest in the newly approve use of XR-NTX for opioid treatment, its effectiveness has not been evaluated in any correctional facilities, including large municipal jails, vs. usual care, nor in the context of standard-of-care methadone treatment. This study will allow providers, correctional and public health authorities, including our collaborators at the NYC Department of Health and Mental Hygiene, and payers and policy makers to assess the utility of XR-NTX as re-entry opioid treatment, with important implications for limiting the great public safety and societal costs of heroin and prescription opioid addictions. Further, NYC jail inmates are predominantly African American and Hispanic, and represent communities disproportionately affected by unemployment, family poverty, HIV and hepatitis C, all downstream effects of opioid dependence. As the majority of opioid addicted persons leave jail return to their neighborhoods untreated and prone to rapid relapse, we hypothesize adding XR-NTX to the re-entry 'toolbox' will save both money and lives in these under-served communities.

This study is part of the NIDA "Studies of Medication for Addiction Treatment in Correctional Settings (SOMATICS)" U01 Collaborative. Our distinct NIH-funded study at NYU has been aligned with two other jail-based opioid treatment studies conducted by researchers at Friends Research Institute (FRI) in Baltimore, MD, and at UCLA. SOMATICS seeks to harmonize assessments and interventions across the three research centers (RCs) and the three independent studies in order to leverage power, sample size, and increase the generalizability of findings. Each of the RCs in the SOMATICS cooperative will conduct their own individual trial, sharing one study arm with another RC, and several core assessments across all sites. The SOMATICS collaborative will have a common Statistical Analysis Plan and DSMP including a single DSMB. The collaborative primary and secondary outcomes across all sites are listed below:

Collaborative Primary Outcome Measures:

1. DSM-5 Opioid Use Disorder Diagnosis during the 30 days prior to the 6 months post-release follow-up assessment: Measured by: DSM-5 checklist via a modified CIDI-2 Substance Abuse Module.

Collaborative Secondary Outcome Measures:

1. Illicit Opioid use: measured by urine drug testing results at 6 months post-release
2. Number of days incarcerated: Measured by self-report during the 6 months post-release.
3. HIV risk behavior: Measured by self-report (Drug Risk Assessment Battery [RAB] Needle Use score) at the 6-month post-release follow-up assessment.
4. Number of days of Opioids, Cocaine, Alcohol, Benzodiazepines, and/or IV Drug Use: Measured by Time Line Follow Back at 6 months post-release follow-up (TLFB; NYU, UCLA) and ASI (FRI).
5. Non-opioid drug use (Cocaine, Amphetamines, and Benzodiazepines): measured by urine drug testing at 6 months post-release
6. Number of days in any drug abuse treatment: Measured by self-report at 6 months post-release.
7. Number of arrests: Measured by self-report data collected at 6 months post-release.
8. Craving scores (for NYU and UCLA sites only): Measured by self-report craving scale at 6 months post-release.
9. Non-lethal overdose (Yes/No): Measured by self-report during the 6 months post-release.
10. Lethal overdose (Yes/No): Measured by public records data reviewed at 6 months post-release.
11. WHO Quality of Life-BREF (WHOQOL-BREF) score: Measured by self-report at 6 months post-release.
12. Analyses of above same secondary outcomes at 12 months follow-up.
13. Analyses of above same secondary outcomes at 24 months follow-up.

ELIGIBILITY:
Due to the nature of this study, which includes both randomized arms (XR-NTX and enhanced TAU) as well as a non-randomized observational arm (methadone treatment group, MTP) there are separate Inclusion/Exclusion criteria for those randomized vs. Non-Randomized, detailed below.

Randomized Arms (XR-NTX, ETAU)

Inclusion Criteria:

1. Adults >18yo incarcerated in NYC jails with known release dates.
2. DSM-V criteria for current opioid use disorder (DSM-IV opioid dependence).
3. Not currently in or planning to pursue agonist (methadone, buprenorphine) treatment at release.
4. Currently opioid free by history ('detoxed') and with a negative urine for all opioids.
5. General good health as determined by medical evaluation.

Exclusion Criteria:

1. Pregnancy, lactation, or planning conception.
2. Active medical illness (i.e., severe liver disease, congestive heart failure) precluding safe participation.
3. Untreated or poorly controlled psychiatric disorder precluding safe participation.
4. History of allergic reaction to naltrexone.
5. Current chronic pain condition treated with opioids.

Non-Randomized Arm (MTP) Inclusion Criteria

1. Adults >18yo incarcerated in NYC jails with known release dates.
2. DSM-V criteria for current opioid use disorder (DSM-IV opioid dependence).
3. Currently receiving regular methadone maintenance treatment through KEEP.
4. General good health as determined by medical evaluation.

Exclusion Criteria

1. Pregnancy, lactation, or planning conception.
2. Active medical illness (i.e., severe liver disease, congestive heart failure) precluding safe participation.
3. Untreated or poorly controlled psychiatric disorder precluding safe participation.
4. In community methadone treatment program at the time of most recent arrest.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2020-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Lee, MD MS, Principal Investigator — NYU MEDICAL CENTER
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - NYC Department of Corrections: Rikers Island Jail Facilities, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Velasquez M, Flannery M, Badolato R, Vittitow A, McDonald RD, Tofighi B, Garment AR, Giftos J, Lee JD. Perceptions of extended-release naltrexone, methadone, and buprenorphine treatments following release from jail. Addict Sci Clin Pract. 2019 Oct 1;14(1):37. doi: 10.1186/s13722-019-0166-0. PMID 31570100
- [Derived] McDonald RD, Tofighi B, Laska E, Goldfeld K, Bonilla W, Flannery M, Santana-Correa N, Johnson CW, Leibowitz N, Rotrosen J, Gourevitch MN, Lee JD. Extended-release naltrexone opioid treatment at jail reentry (XOR). Contemp Clin Trials. 2016 Jul;49:57-64. doi: 10.1016/j.cct.2016.05.002. Epub 2016 May 10. PMID 27178765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended-Release Naltrexone (XR-NTX) | Enhanced Treatment As Usual (ETAU) | Methadone Treatment Program (MTP)
Started | 61 | 58 | 79
Completed | 59 | 56 | 0
Not Completed | 2 | 2 | 79
Not completed — Participant not released from jail | 2 | 2 | 0
Not completed — Not included in primary outcome analysis | 0 | 0 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-Release Naltrexone (XR-NTX) | Enhanced Treatment As Usual (ETAU) | Methadone Treatment Program (MTP) | Total
Number analyzed (Participants) | 59 | 56 | 79 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.9) | 43.7 (9.8) | 43.7 (9.7) | 43.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 19 | 32
  Male | 52 | 50 | 60 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 35 | 82
  Not Hispanic or Latino | 34 | 34 | 44 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 29 | 30 | 34 | 93
  White | 21 | 14 | 27 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 12 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 59 | 56 | 79 | 194

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Relapse: XRNTX vs. ETAU Following Release From Jail
Description: Our primary aim is to compare time-to-relapse among participants treated with XR-NTX vs. randomized ETAU following release from jail measured up to 24 weeks by Urine Toxicology results and self-report on the TLFB.
Time Frame: up to 24 weeks
Population: MTP is a quasi-experimental cohort, so no data was collected for this arm. The primary outcome is a comparison between XR-NTX vs. ETAU only.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Extended-Release Naltrexone (XR-NTX) | Enhanced Treatment As Usual (ETAU)
Number analyzed (Participants) | 59 | 56
Weeks | 8.6 (8.7) | 5.9 (7.7)

2. Secondary Outcome: Time-to-relapse: XR-NTX vs. Methadone (MTP) Cohort Following Release From Jail
Description: Our secondary aim is to measure time-to-relapse among XR-NTX vs. the non-randomized observational Methadone (MTP) cohort up to 24 weeks following release from jail and measured by Urine Toxicology results and self-report on the TLFB.
Time Frame: up to 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Community Treatment Retention/Initiation Post-release
Description: Community treatment retention/initiation across all arms post-release using the Economic Form 90.
Time Frame: up to 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Any Drug or Alcohol Misuse
Description: Any opioid, alcohol, or other illicit drug misuse, defined as continuous counts of both days, amount/day, and urine toxicologies for heroin or other illicit opioid and other drug use across all arms up to 24 weeks post-release and measured by Urine Toxicology Results and the TLFB.
Time Frame: up to 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Injection Drug Use and HIV Sexual Risk Factors
Description: Injection drug use and HIV sexual risk factors will be assessed across all arms measured post-release from jail and measured using the Risk Assessment Battery.
Time Frame: up to 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Accidental Drug Overdose and Mortality
Description: Accidental drug overdose and mortality across all arms assessed at each follow-up study visit up to 28 weeks post-release from jail measured by self report on the Opioid-Overdose AE/SAE form.
Time Frame: up to 28 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Re-incarceration and Exploratory Cost-effectiveness
Description: Re-incarceration and exploratory cost-effectiveness will be assessed across all arms up to 24 weeks post-release and measured using self-report on the Arrests and Days Incarcerated form and information received from the NYC DOC Inmate Locator online. Cost-effectiveness will be assessed across all arms and measured by the Economic Form 90.
Time Frame: up to 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Adverse events were solicited by questionnaire
Arm/Group | Extended-Release Naltrexone (XR-NTX) | Enhanced Treatment As Usual (ETAU) | Methadone Treatment Program (MTP)
All-Cause Mortality (participants affected / at risk) | 1/59 | 2/56 | 0/79
Serious Adverse Events (participants affected / at risk) | 8/59 | 9/56 | 10/79
Other Adverse Events (participants affected / at risk) | 0/59 | 0/56 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-Release Naltrexone (XR-NTX) (N=59) | Enhanced Treatment As Usual (ETAU) (N=56) | Methadone Treatment Program (MTP) (N=79)
Opioid Overdose (General disorders) | 1 (1) | 5 (5) | 2 (2)
Fatal Opioid Overdose (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical Event or Procedure (Surgical and medical procedures) | 6 (6) | 2 (2) | 5 (5)
Death, Unknown Cause (General disorders) | 0 (0) | 1 (1) | 0 (0)
Prolonged Hospitalization (General disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT01999946/Prot_SAP_000.pdf